CLINICAL TRIAL: NCT06317168
Title: SIMPLifying Elements of Standardized Automated Office Blood Pressure Measurements (Pilot Study)
Acronym: SIMPLE-AOBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: SIMPLE-AOBP
Record Dates: First submitted 2024-03-11; First posted 2024-03-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure
Keywords: blood pressure measurements

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standardized automated office BP measurements (Active Comparator): BP measured using a highly standardized procedure using a validated office-grade device on a bare arm supported at heart level.
  Interventions: Diagnostic Test: Mean awake ambulatory BP measurements
- Sleeved arm (Active Comparator): BP measured using a highly standardized procedure using a validated office-grade device over a standardized sleeve with the arm supported at heart level.
  Interventions: Diagnostic Test: Mean awake ambulatory BP measurements
- Arm not supported (Active Comparator): BP measured using a highly standardized procedure using a validated office-grade device on a bare arm resting vertically.
  Interventions: Diagnostic Test: Mean awake ambulatory BP measurements
- Non-validated device (Active Comparator): BP measured using a highly standardized procedure using a non-validated home device on a bare arm supported at heart level.
  Interventions: Diagnostic Test: Mean awake ambulatory BP measurements

INTERVENTIONS:
Diagnostic Test: Mean awake ambulatory BP measurements — Results from all four arms will be compared to the mean awake ambulatory BP measured on the same arm and started immediately following completion of the testing protocol.

SUMMARY:
This study aims to assess whether removing single elements of the standardized office BP measurement procedure will affect the accuracy towards the mean awake ambulatory BP. Four arms are planned in a randomized order: 1) full standardized procedure, 2) standardized procedure but with cuff placed on a sleeve, 3) standardized procedure but arm resting vertically, 4) standardized procedure but with non-validated device.

This is a pilot study to inform on the sample size required to perform adequately powered large scale studies.

DETAILED DESCRIPTION:
Accurate and reliable blood pressure (BP) measurements are key for hypertension management. To this regard, all hypertension societies recommend using highly standardized automated oscillometric office BP measurements (AOBP) as a way to minimise measurement biases, enhance reproducibility and allow comparability. The standardized AOBP procedure emphasizes the need to measure BP in a controlled environment with optimal body positioning, the use of an appropriately sized cuff over a bare arm and a clinically validated oscillometric BP devices. It is also recommended to average >2 measurements at 30-60 seconds intervals after several minutes of seated rest alone in a quiet room. As such, important barriers exist to implement standardized AOBP in real-life settings, as this procedure requires time, space and patient mobility.

A 2017 meta-analysis evaluated the impact of several elements of oscillometric and auscultatory BP readings on systolic and diastolic BP levels. It showed that while most components of BP measurements appear to influence BP, the majority of included studies were of relatively low methodological quality (including unstandardized BP measurements, lack of randomisation, auscultatory method, absence or differences in rest periods, single readings, single cuff size) and almost none were compared with th gold-standard BP measurement, i.e average awake ambulatory BP measurements (ABPM). Since, two meta-analyses specifically assessing the effect of attendance during AOBP were published and showed conflicting results. While important components of AOBP (rest period and cuff size) were recently tested using a rigorous methodology, data is still missing for most elements.

Simplifying the AOBP procedure could result in improvements in acceptability and implementation. The need to perform this highly standardized procedure exerts pressure on patients, providers and administrative staff. Indeed, patients need to be properly seated alone in a quiet dedicated room in a chair with an arm rest that need to be adjustable to position the upper arm at heart level. This setup is seldom available apart in highly specialized hypertension clinics. Also, the arm must be bare, which can bring discomfort to patients with the requirement to remove their clothing or roll up the sleeves, which introduces another potential source of inaccuracy due to the tourniquet effect or the inability to completely uncover the upper arm. It can also introduce significant time delays in a clinical setting for less mobile patients. Furthermore, the BP device must be clinically validated for its accuracy. The lack of regulation and the ease of online purchase means many patients may be drawn to purchasing less expensive non-validated devices. While this problem may be more widespread in the home setting, not all office BP measuring devices are validated and recommended by Hypertension Canada.

The primary objective of the SIMPLE-AOBP study is to assess whether foregoing, or simplifying, specific elements of the AOBP procedure affects its accuracy towards the gold-standard mean awake ABPM. This study will employ a rigorous methodology (highly standardized measurements, identical settings and rest periods, randomization, blinded assessment of outcomes, averaged multiple BP measurements) to minimise measurement biases not related to the studies elements. The study will focus on three easily addressable elements: 1) the need the measure BP on a bare arm, 2) the requirement of supporting the arm at heart level and 3) the need to use a validated BP device. This trial will provide important pilot data to help design adequately powered large scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old

Exclusion Criteria:

* Upper arm size outside of cuff range of selected devices (<22 cm or >42 cm)
* Permanent atrial fibrillation
* Known severe aortic stenosis
* Ongoing pregnancy
* Inability or unwillingness to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Difference with mean awake ambulatory systolic BP | at enrollment (time 0)
  Difference between systolic BP measured in each study arm (average of 3 measurements) with the mean awake ambulatory systolic BP

SECONDARY OUTCOMES:
Difference with mean awake ambulatory diastolic BP | at enrollment (time 0)
  Difference between diastolic BP measured in each study arm (average of 3 measurements) with the mean awake ambulatory diastolic BP

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will not be shared (pilot study)